CLINICAL TRIAL: NCT06411132
Title: A Multicenter, Observational Study to Evaluate Corneal Neurosensory Abnormalities in Patients With Sjögren's Dry Eye
Brief Title: Study to Evaluate Corneal Neurosensory Abnormalities in Patients With Sjögren's Dry Eye
Acronym: GEMINAE
Status: Terminated | Type: Observational
Why Stopped: The analyses presented are based on a database lock date of 05 March 2025.The study was prematurely interrupted by Dompé following a review of the database, which determined that an acceptable no. of patients was reached to meet the trial objectives.
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Other Study IDs: DEV0123
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-03

CONDITIONS: Sjögren Syndrome; Dry Eye
Keywords: Observational; Dry Eye; Sjögren's dry eye; Multinational
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Full Analysis set: The full analysis set includes all patients who meet all the inclusion criteria and none of the exclusion criteria at the end of the screening procedure. All the analyses on the primary and secondary endpoints will be provided on this population. The screened population consists of all patients who sign the ICF and are assigned a patient identification number.
  Please note that the sample size may vary depending on feasibility.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Primary Objective

- To assess the proportion of patients with Sjögren's dry eye who demonstrate impaired corneal sensitivity.

Secondary Objectives

* To assess corneal sensitivity via Cochet-Bonnet esthesiometer.
* To assess tear secretion via Schirmer I test.
* To assess Ocular Pain Assessment Survey (OPAS) questionnaire results.

DETAILED DESCRIPTION:
This observational clinical study has been designed to evaluate the proportion of patients with confirmed Sjögren's dry eye who presented with neurosensory abnormalities via demonstration of increased ocular pain and/or a decrease in corneal sensitivity.

A multicenter design allowed for a greater diversity of patient population with Sjögren's dry eye.

The number of sites allowed for quick enrollment and expedited results that helped physicians understand the corneal sensitivity levels in the population of patients with Sjögren's dry eye.

This study design was minimally invasive and might be completed in a single visit provided all qualification criteria were met.

This design reduced the time commitment from patients, thereby reducing barriers for enrollment and participation.

Only one eye (study eye) was analyzed for endpoints; if both eyes qualified for the study, the eye with the worse staining (per National Eye Institute [NEI] scale) was the study eye. If staining was equal between eyes, the right eye was the study eye.

Please note that no safety monitoring was captured, as this was an observational and descriptive study, and no study drug was administered. All testing and procedures conducted in this study were performed consistent with clinical practice standards and should not pose any additional risk to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age at time of screening.
2. Confirmed diagnosis of Sjögren's for a minimum of 3 months before enrollment, as determined by either serologic antibody testing (anti-SSA/anti-SSB) or biopsy of minor salivary glands.
3. Confirmed diagnosis of dry eye for a minimum of 3 months before enrollment, as determined by signs and/or symptom assessment.
4. Fluorescein corneal staining with a cobalt blue light must show punctate corneal fluorescein staining or staining consistent with corneal epithelial damage equivalent or greater than 1 on the NEI scale by dry eye at enrollment.
5. Only patients who satisfy all informed consent requirements were included in the study. The patient and/or his/her legal representative should read, sign, and date the IRB-approved informed consent document before any study-related procedures were performed.
6. Patients should have the ability and willingness to comply with study procedures.

Exclusion Criteria:

1. Inability to speak and understand English sufficiently to understand the nature of the study, to provide written informed consent, and to allow the completion of all study assessments.
2. Presence of active ocular infection (bacterial, viral, protozoal) in either eye, as deemed by the Investigator or confirmed culture.
3. Previous use of OXERVATE® ophthalmic solution.
4. Presence of gross epithelial defect, including a defect with stromal involvement.
5. Any concurrent medical condition that, in the judgment of the Investigator, might interfere with the conduct of the study or confound the interpretation of the study results.
6. Any eyelid abnormalities, such as lagophthalmos, entropion, ectropion, or other neuromuscular abnormalities, that result in prolonged exposure of the corneal surface.
7. Concurrent epithelial corneal disease or dystrophy unrelated to dry eye, such as anterior basement membrane dystrophy.
8. Inability to remove contact lenses for a minimum of 3 hours before corneal sensitivity testing.
9. Inability to discontinue use of all topical ophthalmic treatments for a minimum of 3 hours before corneal sensitivity testing.
10. Inability to suspend use of any neurostimulatory drugs or devices (including but not limited to nasal varenicline, iTear100, etc.) for treating dry eye or increasing tear film for 6 hours before testing.
11. Ocular surgery (including but not limited to laser-assisted in situ keratomileusis, photorefractive keratectomy, tube shunt/trabeculectomy, or cataract surgery) within the last 6 months.
12. History of corneal stromal surgery, including anterior lamellar keratoplasty, deep anterior lamellar keratoplasty, and penetrating keratoplasty.
13. Current participation in another clinical study that might affect corneal sensitivity or tear production.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 182 patients were planned to be included in the study. Due to its early termination, a total of 114 patients were screened and 103 patients were included in the FAS. Eleven patients did not meet the inclusion and/or exclusion criteria. All patients (103 patients) completed the study.
  The screened population consisted of all patients who signed the ICF and were assigned a patient identification number. The full analysis set (FAS) included all patients who met all the inclusion criteria and none of the exclusion criteria at the end of the screening procedure.
  All the analyses on the primary, secondary endpoints are provided on this population (FAS).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with Sjögren's dry eye who demonstrate impaired corneal sensitivity | Visit 1 (Day 1)
  The number and proportion of patients with Sjögren's dry eye who have decreased corneal sensitivity, as determined by Cochet-Bonnet esthesiometer, will be shown with the 95% CI (Wilson method).

SECONDARY OUTCOMES:
Corneal sensitivity, as measured via Cochet-Bonnet esthesiometer. | Visit 1 (Day 1)
  Summary statistics for continuous and categorical variables will be used to assess the secondary endpoints. Any statistical testing will be descriptive in nature.
Tear secretion, as measured via Schirmer I test. | Visit 1 (Day 1)
  Summary statistics for continuous and categorical variables will be used to assess the secondary endpoints. Any statistical testing will be descriptive in nature.
OPAS questionnaire results. | Visit 1 (Day 1)
  Summary statistics for continuous and categorical variables will be used to assess the secondary endpoints. Any statistical testing will be descriptive in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hauswirth, OD, Study Director — Dompé Farmaceutici SpA
Locations (15):
- United States (15):
  - West Coast Eye Institute, Bakersfield, California
  - University of Colorado, Aurora, Colorado
  - Bowden Eye, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - Minnesota Eye Consultants, Woodbury, Minnesota
  - Eye Associates of North Jersey, Dover, New Jersey
  - Weil Cornell Medicine, New York, New York
  - Triangle Eye Consultants, Raleigh, North Carolina
  - Vita Eye Clinic, Shelby, North Carolina
  - Focus Eye Care, Wilmington, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Toyos Clinic, Nashville, Tennessee
  - Periman Eye Institute, Seattle, Washington